CLINICAL TRIAL: NCT02806713
Title: The Effect of Oral phenazopyrIdine on Perioperative Voiding After Mid-urethral Sling
Brief Title: The Effect of Oral PhenazopyrIdine on Perioperative Voiding After Mid-urethral sliNg (EPIPhANy Study)
Acronym: EPIPhANy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Michael Flynn, Principal Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H00008816
Record Dates: First submitted 2016-04-29; First posted 2016-06-21 (Estimated); Results first posted 2019-02-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-01

CONDITIONS: Dysfunctional Voiding; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Phenazopyridine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- no phenazopyridine (Placebo Comparator): Patients not receiving phenazopyridine (standard of care)
  Interventions: Other: no Phenazopyridine
- phenazopyridine (Experimental): Patients receiving phenazopyridine
  Interventions: Drug: Phenazopyridine

INTERVENTIONS:
Drug: Phenazopyridine
  Other Names: Pyridium
  Arms: phenazopyridine
Other: no Phenazopyridine — Because the obvious effects on the urine coloration of pyridium no placebo or dummy are provided
  Arms: no phenazopyridine

SUMMARY:
Randomized clinical trial using phenazopyridine to decrease voiding dysfunction after a retropubic midurethral sling operation.

DETAILED DESCRIPTION:
Study design and randomization This study is a randomized controlled trial. Randomization will be performed using software and a block randomization scheme. Study assignment will be completed using sequentially numbered sealed opaque envelopes. All the research procedures described other than the use or not of phenazopyridine will be applicable to both arms of the study. Subjects will have a 50% chances of getting either phenazopyridine or nothing.

Because pyridium turns the urine orange, it is impossible to blind the patients and researchers to the study assignment. Because there is no known placebo that turns the urine orange, there is no value to using an actual placebo tablet. Subjects will be assigned to either receive pyridium or not receive pyridium preoperatively.

Screening potential subjects: Investigators will screen potential subjects for contraindications to methylene blue. Prior obtaining the routine surgical consent for the potential subject's surgical procedure, the patient's medical history in the UMass Electronic Medical Record is routinely reviewed. The medical record will be reviewed for a diagnosis of G6PD and if found, the potential subject will be excluded.

Once written consent has been obtained, subject number will be assigned and the appropriate randomization envelope will be opened. The study assignment will not be formally shared with the subject. Those assigned to the "pyridium" arm will have orders written for the standard 200 mg dose of pyridium to be given on arrival to the Surgical Admissions Care Unit (SACU). Those assigned to the "NO pyridium" arm with have their routine preoperative orders written along with an order for "No preoperative pyridium".

Subjects will then follow the routine perioperative care for their procedures with the only study interventions being the gathering of PHI and performing postoperative pain assessments.

PHI will be obtained at the time of the surgical consent with the purpose to evaluate for possible confounders affecting the postoperative bladder function.

Surgical procedure:

The Mid Urethral Sling will be performed in standard fashion based on manufacturer's recommendations and instructions to minimize inter-observer variations. We will perform the procedure according to our usual and customary techniques. The subject will receive the same technique and interventions that a routine patient on the Urogyn service would expect to undergo. There will be no changes to the technique for the purpose of the study.

Bladder challenge:

Patient will undergo voiding trial at same day surgery per our usual and customary protocol. This is the same protocol the subject would undergo as a patient on the Urogyn service. The bladder challenge will be interpreted in our usual manner and the subject managed according to our routine clinical protocols.

Postoperative care:

Subjects will undergo routine postoperative care and followup. Subjects failing their bladder challenge will be seen in the Urogyn clinic according to routine clinical protocols and data concerning their void trials collected. Subjects will undergo routine followup evaluation 6 weeks postoperatively in the order to assess any potential long-term voiding dysfunction. Information on any postoperative complications will be collected

Administration of Visual analog scale:

(1) Visual analog scale for assessment of pain will be administered at two- time intervals.

1. VAS #1) Preoperative VAS will be done by the principal investigator or any of the study assistants. The VAS form will be part of subject's packet.
2. VAS#2) VAS will be administered by one of the study investigators 2 to 3 hours after the surgical procedure in the SACU.

ELIGIBILITY:
Inclusion Criteria:

1. Any female subjects scheduled to undergo Mid-Urethral Sling (MUS) through the UMass urogynecology service for incontinence.

Exclusion Criteria:

1. Planned concurrent prolapse or other procedure besides cystoscopy
2. Using intermittent self catheterization preoperatively
3. Undergoing spinal anesthesia for the procedure
4. Known allergy to phenazopyridine (AKA Pyridium)
5. Renal insufficiency
6. Any condition or situation that in the attending physician's opinion would contra-indicate the use of phenazopyridine
7. Subjects not competent to give consent
8. Prisoners
9. Non-English speaking patients
10. Age <18
11. Pregnant patients
12. Contraindications to the use of IV methylene blue including

    1. Patients with known hypersensitivity reactions
    2. Severe renal insufficiency
    3. Patients with G6PD deficiency

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2016-02; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael K Flynn, MD, MHS, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- Umass Memorial, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nilsson CG, Kuuva N, Falconer C, Rezapour M, Ulmsten U. Long-term results of the tension-free vaginal tape (TVT) procedure for surgical treatment of female stress urinary incontinence. Int Urogynecol J Pelvic Floor Dysfunct. 2001;12 Suppl 2:S5-8. doi: 10.1007/s001920170003. PMID 11450979
- [Background] Nilsson CG, Palva K, Rezapour M, Falconer C. Eleven years prospective follow-up of the tension-free vaginal tape procedure for treatment of stress urinary incontinence. Int Urogynecol J Pelvic Floor Dysfunct. 2008 Aug;19(8):1043-7. doi: 10.1007/s00192-008-0666-z. Epub 2008 Jun 6. PMID 18535753

RESULTS

PARTICIPANT FLOW:
Groups:
- Phenazopyridine: Patients receiving phenazopyridine
  Phenazopyridine
Period: Overall Study
Arm/Group | no Phenazopyridine | Phenazopyridine
Started | 46 | 46
Completed | 44 | 44
Not Completed | 2 | 2
Not completed — Urethral injury during procedure | 1 | 0
Not completed — cancelled surgery | 1 | 2

BASELINE CHARACTERISTICS:
Population: we started with 46 subjects per arm, 2 cancelled surgery and 1 had an intraoperative urethral injury.
Groups:
- Total: Total of all reporting groups
Arm/Group | no Phenazopyridine | Phenazopyridine | Total
Number analyzed (Participants) | 44 | 44 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 44 | 44 | 88
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (9.4) | 49.7 (12.6) | 48.7 (11.1)
Age, Continuous [Mean (Full Range); unit: years] | 47.7 [35 to 68] | 49.7 [37 to 61] | 48.7 [35 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 44 | 88
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 8 | 13
  Not Hispanic or Latino | 39 | 36 | 75
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 33 | 29 | 62
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 9 | 18
Region of Enrollment [Number; unit: participants]
  United States | 44 | 44 | 88

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Failed Voiding Trial
Description: Number of participants with a failed postoperative voiding trial. A failed voiding trial is defined as not voiding all urine in 20 minutes or voiding less than 1/3 of total volume (voided volume + post void residual). Patients will undergo voiding trial at same day surgery per the following protocol. Participants who do not pass the voiding trial the same day of their surgical procedure return to the clinic in 3 days to repeat it, following the same protocol described above.
Time Frame: Postoperatively, up to 3 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | no Phenazopyridine | Phenazopyridine
Number analyzed (Participants) | 44 | 44
Participants
  Passed the voiding trial | 35 | 32
  Failed a voiding trial | 9 | 12

2. Secondary Outcome: Change in Participant-reported Pain From Pre to Post Procedure Using the Visual Analog Scale (VAS)
Description: To determine if the phenazopyridine has an analgesic effect after the retropubic midurethral slings, participants will be asked to self-report pain intensity preoperatively and then postoperatively (2 to 3 hours post procedure) using the Visual Analog Scale (VAS). The scale of the VAS is from 0 meaning "no pain" to 10 indicating the "worst pain." The resulting change is measured as the difference between the self-reported preoperative pain score and the postoperative pain score.
Time Frame: Preoperatively and then 2 to 3 hours after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | no Phenazopyridine | Phenazopyridine
Number analyzed (Participants) | 44 | 44
score on a scale | 1.76 (1.31) | 1.21 (1.2)

ADVERSE EVENTS:
Time Frame: Up to six weeks postoperatively
Arm/Group | no Phenazopyridine | Phenazopyridine
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 0/44 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-07): https://cdn.clinicaltrials.gov/large-docs/13/NCT02806713/Prot_SAP_000.pdf